CLINICAL TRIAL: NCT02767271
Title: An Open-Label Study to Assess the Pharmacokinetics With Maximal Use of Luliconazole Cream 1% in Pediatric Patients With Moderate to Severe Tinea Pedis or Tinea Cruris
Brief Title: Maximal Use of Luliconazole Cream 1% in Pediatric Participants With Moderate to Severe Tinea Pedis or Tinea Cruris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V01-LUZA-401
Record Dates: First submitted 2016-05-03; First posted 2016-05-10 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Tinea Pedis; Tinea Cruris
MeSH Terms: conditions — Tinea Pedis; Tinea Cruris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tinea Pedis (Experimental): Participants with tinea pedis received luliconazole cream 1% topically once daily in the morning for 15 days (Day 1 through 15). The dose was approximately 3.0 grams per application and covered all affected and adjacent areas, including up to the ankles.
  Interventions: Drug: Luliconazole Cream 1%
- Tinea Cruris (Experimental): Participants with tinea cruris received luliconazole cream 1% topically once daily in the morning for 8 days (Day 1 through 8). The dose was approximately 3.0 grams per application and covered all affected and adjacent areas, including up to the groin, thighs, and abdomen.
  Interventions: Drug: Luliconazole Cream 1%

INTERVENTIONS:
Drug: Luliconazole Cream 1% — Luliconazole cream will be applied topically per schedule specified in the arms.

SUMMARY:
The objective of this study is to evaluate the pharmacokinetics of luliconazole cream 1%, as measured by circulating plasma levels of luliconazole, when maximal quantity of luliconazole cream 1% is applied to participants of 12 years to less than (<) 18 years of age with moderate to severe inter-digital tinea pedis or tinea cruris.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants (or legal guardian) with the ability and willingness to sign a written informed consent.
* Participants of either gender at least 12 years to <18 years old (12 to 17 years, inclusive).
* Participants with a mycological diagnosis of tinea pedis or tinea cruris confirmed by the detection of fungal hyphae on a microscopic potassium hydroxide (KOH) wet mount.
* Participants with the ability and willingness to follow all study procedures, attend all scheduled visits, have all blood draws, and successfully complete the study.
* Participants must be in good general health and free of any disease that in the Investigator's opinion might interfere with the study evaluations.
* Participants must be able to communicate, be able to understand the study procedures, and be willing to comply with the study requirements.

Key Exclusion Criteria:

* Participants with both tinea pedis and tinea cruris.
* Participants with active atopic or contact dermatitis in the treatment area.
* Female participants who are pregnant and/or nursing or planning a pregnancy during the course of the trial. Participants who test positive for pregnancy after start of test treatment will be discontinued from test treatment but will be followed for safety purposes.
* Participants who are immunocompromised (due to disease, for example; human immunodeficiency virus [HIV] or medications).
* Participants who have a recent history of or current drug or alcohol abuse.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2016-04-27 (Actual); Study Completion 2016-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Valeant Pharmaceuticals
Locations (2):
- Valeant Site 01, Santo Domingo, Dominican Republic
- Valeant Site 02, San Pedro Sula, Honduras

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tinea Pedis: Participants with tinea pedis received luliconazole cream 1% topically once daily in the morning for 15 days (Day 1 through 15). The dose was approximately 3.0 grams per application and covered all affected and adjacent areas.
- Tinea Cruris: Participants with tinea cruris received luliconazole cream 1% topically once daily in the morning for 8 days (Day 1 through 8). The dose was approximately 3.0 grams per application and covered all affected and adjacent areas.
Period: Overall Study
Arm/Group | Tinea Pedis | Tinea Cruris
Started | 15 | 15
Safety Population (Received at least 1 application of study drug.) | 15 | 15
Pharmacokinetic Pedis (PKP) Population (Participants with tinea pedis, received ≥1 dose of study drug, had at least 1 PK assessment.) | 15 | 0
Pharmacokinetic Cruris (PKC) Population (Participants with tinea cruris, received ≥1 dose of study drug, had at least 1 PK assessment.) | 0 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were enrolled and received at least 1 application of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tinea Pedis | Tinea Cruris | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.13 (2.17) | 15.27 (1.49) | 14.70 (1.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Circulating Plasma Levels of Luliconazole in Participants Who Had Tinea Pedis: Maximum Observed Plasma Concentration (Cmax) of Luliconazole
Description: Plasma concentration of luliconazole was determined using validated liquid chromatography-mass spectrometry (LC/MS) method.
Time Frame: Pre-dose (15 minutes) and at 1, 3, 6, 9, 12, and 24 hours post-dose on Day 15
Population: PKP population included all participants with tinea pedis who were enrolled, received at least 1 application of study drug, and had at least 1 pharmacokinetic (PK) assessment.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Tinea Pedis
Number analyzed (Participants) | 15
nanograms/milliliter (ng/mL) | 3.27 (1.71)

2. Primary Outcome: Measurement of Circulating Plasma Levels of Luliconazole in Participants Who Had Tinea Pedis: Area Under the Plasma Concentration Versus Time Curve From Time 0 to 24 Hours (AUC0-24) of Luliconazole
Description: Plasma concentration of luliconazole was determined using validated LC/MS method. AUC0-24 was calculated by linear trapezoidal method.
Time Frame: Pre-dose (15 minutes) and at 1, 3, 6, 9, 12, and 24 hours post-dose on Day 15
Population: PKP population included all participants with tinea pedis who were enrolled, received at least 1 application of study drug, and had at least 1 PK assessment.
Measure: Mean (Standard Deviation); unit: nanograms*hour/milliliter (ng*hr/mL)
Arm/Group | Tinea Pedis
Number analyzed (Participants) | 15
nanograms*hour/milliliter (ng*hr/mL) | 60.38 (37.92)

3. Primary Outcome: Measurement of Circulating Plasma Levels of Luliconazole in Participants Who Had Tinea Pedis: Elimination Half-Life (t1/2) of Luliconazole
Description: Plasma concentration of luliconazole was determined using validated LC/MS method.
Time Frame: Pre-dose (15 minutes) and at 1, 3, 6, 9, 12, and 24 hours post-dose on Day 15
Population: PKP population included all participants with tinea pedis who were enrolled, received at least 1 application of study drug, and had at least 1 PK assessment. None of the participants in this population was evaluable for this outcome measure at specified timepoint.
Arm/Group | Tinea Pedis
Number analyzed (Participants) | 0

4. Primary Outcome: Measurement of Circulating Plasma Levels of Luliconazole in Participants Who Had Tinea Cruris: Cmax of Luliconazole
Description: Plasma concentration of luliconazole was determined using validated LC/MS method.
Time Frame: Pre-dose (15 minutes) and at 1, 3, 6, 9, 12, and 24 hours post-dose on Day 8
Population: PKC population included all participants with tinea cruris who were enrolled, received at least 1 application of study drug, and had at least 1 PK assessment.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tinea Cruris
Number analyzed (Participants) | 15
ng/mL | 15.40 (13.62)

5. Primary Outcome: Measurement of Circulating Plasma Levels of Luliconazole in Participants Who Had Tinea Cruris: AUC0-24 of Luliconazole
Description: as for outcome 2
Time Frame: Pre-dose (15 minutes) and at 1, 3, 6, 9, 12, and 24 hours post-dose on Day 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Tinea Cruris
Number analyzed (Participants) | 15
ng*hr/mL | 266.06 (236.07)

6. Primary Outcome: Measurement of Circulating Plasma Levels of Luliconazole in Participants Who Had Tinea Cruris: t1/2 of Luliconazole
Description: Plasma concentration of luliconazole was determined using validated LC/MS method.
Time Frame: Pre-dose (15 minutes) and at 1, 3, 6, 9, 12, and 24 hours post-dose on Day 8
Population: PKC population included all participants with tinea cruris who were enrolled, received at least 1 application of study drug, and had at least 1 PK assessment. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tinea Cruris
Number analyzed (Participants) | 3
hours | 49.77 (22.74)

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to Day 16
Description: Safety population included all participants who were enrolled and received at least 1 application of study drug.
Arm/Group | Tinea Pedis | Tinea Cruris
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 2/15 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tinea Pedis (N=15) | Tinea Cruris (N=15)
Diarrhea (Gastrointestinal disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.